CLINICAL TRIAL: NCT00051441
Title: A Double-Blind, Randomized, Vehicle-Controlled Study Comparing the Safety and Efficacy of Benzydamine HCl 0.15% Oral Rinse Including a Separate Open-Label Standard of Care Arm in Subjects With Radiation-Induced Mucositis
Brief Title: Safety & Efficacy Study of Benzydamine Oral Rinse for the Treatment of Oral Mucositis (Mouth Sores) Resulting From Radiation Therapy for Cancer of the Oral Cavity, Oropharynx, or Nasopharynx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Collaborators: Angelini (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002491
Record Dates: First submitted 2003-01-09; First posted 2003-01-13 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Stomatitis; Radiation Effects
Keywords: stomatitis; radiation effects
MeSH Terms: conditions — Stomatitis | interventions — Benzydamine; Mouthwashes

INTERVENTIONS:
Drug: Benzydamine Hydrochloride 0.15% Oral Rinse

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of benzydamine hydrochloride 0.15% oral rinse to a vehicle oral rinse in the treatment of radiation-induced oral mucositis, and to compare the care normally used for radiation-induced oral mucositis to vehicle oral rinse to ensure that the vehicle does not have detrimental effects on the oral mucosa

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, vehicle-controlled study including an open-label standard of care arm, to determine the effectiveness and safety of benezydamine hydrochloride 0.15% oral rinse as compared with vehicle oral rinse, and vehicle oral rinse as compared to the care normally used in the treatment of radiation-induced oral mucositis. The hypotheses are that benzydamine hydrochloride 0.15% oral rinse is better than vehicle oral rinse as measured by the proportion of patients reaching a WHO mucositis score of 3 by 5500 cGy and vehicle is no worse than the standard of care as measured by the proportion of patients reaching a WHO mucositis score of 3 by 5500 cGy. Patients receiving benzydamine hydrochloride 0.15% or vehicle double-blind oral rinses will place 15 mL in the mouth for 2 minutes, gargling for a few seconds at the beginning and end of the rinse, and then expectorate the entire dose. Dosing with oral rinses will be every 2 - 3 hours while awake for a minimum of 4 times daily to a maximum of 8 times per day. Double-blind oral rinses will continue daily throughout the duration of the subjects radiation treatment regimen plus 2 additional weeks

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance scale >= 60%
* Diagnosis of pathologically confirmed malignancy involving one or more of the following sites: oral cavity, oropharynx extending down to the level of the supraglottic area, nasopharynx, maxillary sinus and parotid gland
* high risk for developing oral and/or oropharyngeal mucositis due to radiation to head and neck areas
* scheduled to receive a continuous course (eg, often six to eight weeks) of conventional or hyperfractionated external beam radiation for cancer of the head and neck region (subjects who had surgery prior to radiation are eligible) with or without concomitant chemotherapy
* at least two oral tissue sites (not including areas of previous lesions, tumor, surgical resection, or the lips) must be included in the RT treatment volume and planned to receive a total radiation dose of 5500 cGy or higher, given in a single daily fraction of 180 to 220 cGy or twice daily fractions of 110 to 150 cGy

Exclusion Criteria:

* Known hypersensitivity to benzydamine HCl and/or any of the other components including alcohol, menthol, glycerin, flavoring agents, and preservatives
* oral or oropharyngeal mucositis present at the time of entry into the study
* treatment regimen consisting of noncontinuous radiation therapy
* received chemotherapy within 21 days of entry into the study as defined by initiation of radiation
* scheduled to receive or have received brachytherapy
* chronically being medicated for conditions other than tumor-related pain with oral and/or parenteral prescription steroids or analgesics
* use of chlorhexidine gluconate (Peridex), amifostine (Ethyol), topical antibiotics to the mouth (ie, tetracycline), topical steroids to the mouth, povidone iodine rinses, glutamine oral rinses, selective decontamination, and Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF)
* use of mouthwash containing other exclusionary medications and any other medication(s) without an approved indication for topical oral use with the exception of liquid antacid formulations (eg, Maalox, Mylanta)
* participated in an investigational study within 30 days prior to enrolling into the study where an experimental drug and/or product was taken
* not willing and/or able to take opioids for any reason
* cryotherapy (ie, ice chips or popsicles) prior to or during chemotherapy infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the cumulative proportion of patients with severe mucositis (WHO mucositis score of at least 3) at a cumulative radiation dose of 5500 cGy

SECONDARY OUTCOMES:
Secondary endpoints include cumulative RT to first use of an opioid for oral mucositis; cumulative RT to first ulceration; cumulative RT to first RT suspension due to oral mucositis

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: Safety and Efficacy Study of Benzydamine Oral Rinse for the Treatment of Oral Mucositis (Mouth Sores) Resulting From Radiation Therapy for Cancer of the Oral Cavity, Oropharynx, or Nasopharynx — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=904&filename=CR002491_CSR.pdf